CLINICAL TRIAL: NCT03304366
Title: The Use of Pentacam in Assessment of Corneal Changes After Pterygium Excision
Brief Title: Corneal Changes With Pentacam Before and After Pterygium
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal, Resident Physician, Assiut University
Other Study IDs: Pentacam
Record Dates: First submitted 2017-10-04; First posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with primary pterygium: * All eyes have primary pterygium and seeking for surgery due to Cosmetic problems, ocular irritation, and, or visual impairment.
  * All selected patients will undergo complete ophthalmological examination including refraction, best corrected visual acuity, keratometry, and pentacam (scheimpflug imaging) preoperatively then will be followed up 2 and 6 months post pterygium excision.
  Interventions: Diagnostic Test: Pentacam (scheimpflug imaging)

INTERVENTIONS:
Diagnostic Test: Pentacam (scheimpflug imaging) — Corneal changes including thickness, elevations....etc

SUMMARY:
Aim of this study is to assess the corneal changes before and after pterygium excision by using pentacam system.

DETAILED DESCRIPTION:
Pterygium is a dysplasia of the bulbar conjunctiva extending onto the corneal surface. The prevelance of pterygium ranges from 0.7% to 31% in various populations according to the location, altitude, and race. It has a higher prevelance in areas which have increased exposure to direct sun with ultraviolet (UV) B light. Patients with pterygia present with variety of complaints ,ranging from asymptomatic to significant redness ,swelling ,itching ,irritation and blurring of vision associated with elevated lesions of the conjunctiva and contiguous cornea in one or both eyes.The induction of astigmatism due to the invasion of the pterygium into the cornea as well as changes in corneal curvature and refractive status has been reported by numerous studies.

Multiple different procedures have been advocated in the treatment of pterygia. These procedures range from simple excision to sliding flaps of conjunctiva with or without adjunctive external beta radiation therapy and/or use of topical chemotherapeutic agents, such as Mitomycin C.

Pentacam is a rotating Scheimpflug camera which measures Scheimpflug images of the anterior eye segment. With the pentacam, topographic analysis of the corneal front and back surfaces is based on the true elevation measurement from one side of the cornea to the other (limbus to limbus). Pentacam also describes the true thickness of the cornea across its entire breadth and width.

Type of the study: prospective observational longitudinal study

Study Setting: Assuit University Hospital ( ophthalmology Department ) Assuit Police Hospital ( ophthalmology Department )

Study subjects:

1. Inclusion criteria:

   * The study will include 30 eyes of adult subjects.
   * All eyes have primary pterygium and seeking for surgery due to Cosmetic problems, ocular irritation, and, or visual impairment.
   * All selected patients will undergo complete ophthalmological examination including refraction, best corrected visual acuity, keratometry, and pentacam (scheimpflug imaging) preoperatively then will be followed up 2 and 6 months post pterygium excision.
2. Exclusion criteria:

   * patients with recurrent pterygium.
   * Patients with media opacities:

     * Dense cataract. - Corneal opacities.
   * Patients with a history of intraocular surgery ,ocular trauma ,and contact lens wear.
   * Patients with severe ocular surface disorders as Stevens-Johnson syndrome.

ELIGIBILITY:
Inclusion Criteria:

* All eyes have primary pterygium and seeking for surgery due to Cosmetic problems, ocular irritation, and, or visual impairment.
* All selected patients will undergo complete ophthalmological examination including refraction, best corrected visual acuity, keratometry, and pentacam (scheimpflug imaging) preoperatively then will be followed up 2 and 6 months post pterygium excision.

Exclusion Criteria:

* patients with recurrent pterygium.
* Patients with media opacities: Dense cataract, Corneal opacities.
* Patients with a history of intraocular surgery ,ocular trauma ,and contact lens wear.
* Patients with severe ocular surface disorders as Stevens-Johnson syndrome.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary pterygium comes to Assiut University Hospital, Assiut Police Hospital, Private clinic They will perform the Pentacam analysis at Assuit Eye research centers (Alforsan-Elnoor)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Pentacam analysis. | preoperative and then will be followed up 2 and 6 months post pterygium excision.
  Corneal changes such as thickness and elevations

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S Abdelrahman, Prof, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided
Sharing the results for other researchers